CLINICAL TRIAL: NCT01046175
Title: Effect of Two Different Air-stacking Techniques, Combined With Manually Assisted Cough, on Peak Cough Flow (PCF) in Patients With Acute Cervical or High Thoracic Spinal Cord Injury
Brief Title: Effect of Air-stacking on Peak Cough Flow in Patients With Acute Cervical or High Thoracic Spinal Cord Injury
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of patients. Investigator changed job.
Sponsor: Ullevaal University Hospital (Other)
Responsible Party: Post doc research fellow Helene L. Soberg, Oslo University Hospital, Ullevaal, Dept. of Phys. Med & Rehab.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: S-09326b
Record Dates: First submitted 2009-12-22; First posted 2010-01-11 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2009-12

CONDITIONS: Spinal Cord Injury; Tetraplegia
Keywords: Respiratory complications; respiratory insufficiency; respiratory therapy
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia; Respiratory Insufficiency | interventions — Ventilators, Mechanical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Airstacking with manual resuscitator (Experimental): Air-stacking is a type of lung volume recruitment technique where insufflations are stacked in the lungs to maximally expand them, here done with a manual resuscitator.
  Interventions: Procedure: Air-stacking with a manual resuscitator
- Air-stacking with ventilator (Active Comparator): Air-stacking is a type of lung volume recruitment technique where insufflations are stacked in the lungs to maximally expand them, here done with a ventilator.
  Interventions: Procedure: Air-stacking with ventilator

INTERVENTIONS:
Procedure: Air-stacking with a manual resuscitator — Stacking air into the lungs up to maximal insufflation capacity (MIC)with a manual resuscitator
  Other Names: Lung volume recruitment technique
  Arms: Airstacking with manual resuscitator
Procedure: Air-stacking with ventilator — Stacking air into the lungs to maximal insufflation capacity (MIC) with ventilator
  Other Names: Lung volume recruitment technique
  Arms: Air-stacking with ventilator

SUMMARY:
Respiratory complications continue to be one of the leading causes of morbidity and mortality in people with spinal cord injury, especially among cervical and higher thoracic injuries. Both inspiratory and expiratory function are often severely decreased, leading to respiratory complications, such as atelectasis, pneumonia and ventilatory failure. The prevention of these respiratory complications needs to begin immediately after injury. To achieve effective expelling of secretions before they form mucus plugs, it is essential to improve patients ability to cough. Manually assisting the cough is one way of increasing cough flow, but an effective cough also requires adequate lung volumes. The emphasis should therefore be on expansion of the lungs before coughing. One way of expanding the lungs is by air-stacking. In air-stacking insufflations are stacked in the lungs to maximally expand them. Cough can be valued by measuring Peak Cough Flow (PCF). By combining air-stacking with manually assisted cough the PCF can be increased sufficiently. The aim of this study is to compare the effect of two different air-stacking techniques on PCF, air-stacking on a respirator versus air-stacking with a manual resuscitator.

ELIGIBILITY:
Inclusion Criteria:

* acute cervical or high thoracic spinal cord injury admitted to the ICU

Exclusion Criteria:

* substantial abdominal or thoracic injury
* substantial brain damage
* intubated or tracheostomized patients
* not able to cooperate
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-02 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Peak cough flow (PCF) | 2 weeks

SECONDARY OUTCOMES:
Patient preference of air-stacking technique | 2 weeks
Physiotherapist preference of air-stacking technique | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Helene L Soberg, PhD, Study Chair — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Ullevaal, Oslo, Norway